CLINICAL TRIAL: NCT04462952
Title: A Phase I, Open-label Study to Assess the Safety, Tolerability, Pharmacokinetics and Anti-Tumour Activity of Adavosertib (AZD1775) in Monotherapy and in Combination With Chemotherapy in Japanese Patients With Advanced Solid Tumours
Brief Title: Study of Adavosertib(AZD1775) in Japanese Patients With Advanced Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D601HC00008
Record Dates: First submitted 2020-06-17; First posted 2020-07-08 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Advanced Solid Tumours
MeSH Terms: interventions — adavosertib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adavosertib (AZD1775) monotherapy (Experimental): Dose escalation of adavosertib monotherapy for patients with advanced solid tumours
  Interventions: Drug: Adavosertib (AZD1775)
- Adavosertib (AZD1775) in combination with gemcitabine (Experimental): Dose escalation of adavosertib in combination with gemcitabine for patients with advanced solid tumours
  Interventions: Drug: Adavosertib (AZD1775)

INTERVENTIONS:
Drug: Adavosertib (AZD1775) — Adavosertib taken orally

SUMMARY:
This is a phase I, open-label study to assess the safety, tolerability, pharmacokinetics(PK) and anti-tumour activity of adavosertib in Japanese patients with advanced solid tumours. This study consists of 2 parts, monotherapy (part A) and chemotherapy combination (part B). At least 3, or up to 6, evaluable Japanese patients with advanced solid tumours will be enrolled in each cohort to confirm the tolerability.

DETAILED DESCRIPTION:
Objectives:

Primary objective:

Part A:

To assess the safety and tolerability, describe any dose-limiting toxicity (DLT) for adavosertib

Secondary objective:

To determine the PK profile of adavosertib To describe adavosertib's preliminary anti-tumour activity using the Response Evaluation Criteria in Solid Tumours (RECIST) v1.1

Part B:

To assess the safety and tolerability, describe any dose-limiting toxicity (DLT) for adavosertib in combination with gemcitabine

Secondary objective:

To determine the PK profile of adavosertib plus gemcitabine To describe preliminary anti-tumour activity of adavosertib in combination with gemcitabine using the Response Evaluation Criteria in Solid Tumours (RECIST) v1.1 To assess the drug interaction between adavosertib and gemcitabine

Overall design:

This is a phase I, open-label study to assess the safety, tolerability, PK and anti-tumour activity of adavosertib in Japanese patients with advanced solid tumours. This study consists of 2 parts, monotherapy (part A) and chemotherapy combination (part B). At least 3, or up to 6, evaluable Japanese patients with advanced solid tumours will be enrolled in each cohort. The total number of subjects will depend upon the available data in each cohort and the Safety Review Committee (SRC)'s decision.

Number of Subjects:

At least 3, or up to 6, evaluable Japanese patients with advanced solid tumours will be enrolled in each cohort.

Treatments and treatment duration:

Subjects in each part will receive the study treatments as described below:

Part A: Adavosertib by mouth (PO) once daily (QD) for 5 days ON and 2 days OFF for week 1 and 2 of a 21 days cycle.

Part B: Adavosertib PO will be taken QD on Days 2, 3, 9, 10, 16, and 17. Gemcitabine will be administered by intravenous infusion according to institutional standards on Days 1, 8, and 15 of each 28-day cycle.

Subjects will be allowed to continue adavosertib until disease progression, intolerable toxicity, or discontinuation criteria have been met.

ELIGIBILITY:
Major Inclusion Criteria:

* Japanese patients ≥20 years of age at the time of study entry
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0, 1
* Adequate bone marrow reserve or organ function
* Female patients who are not of child-bearing potential, and fertile females of childbearing potential who agree to use adequate contraceptive measures
* Male patients should be willing to use barrier contraception
* Predicted life expectancy ≥12 weeks
* Part A : Histologically or cytologically documented locally advanced or metastatic solid tumour, excluding lymphoma, for which standard therapy does not exist or has proven ineffective or intolerable
* Part B : Histologically or cytologically documented locally advanced or metastatic solid tumour, excluding lymphoma, for which standard therapy does not exist or has proven ineffective or intolerable and additionally, tumours for which gemcitabine is expected to be effective.
* Measurable or non-measurable disease according to RECIST v1.1

Major Exclusion Criteria:

* Use of anti-cancer treatment drug ≤21 days or 5 half-lives (whichever is shorter) prior to Cycle 1 Day 1
* Use of an investigational drug during the past 30 days or 5 half-lives (whichever is longer) prior to Cycle 1 Day 1
* Common Terminology Criteria for Adverse Events (CTCAE) Grade >1 toxicity from prior therapy
* Inability to swallow oral medication or any other condition that may impact adavosertib intake/absorption
* Known malignant central nervous system (CNS) disease other than neurologically stable, treated brain metastases
* Any of the cardiac diseases currently or within the last 6 months
* Any underlying medical condition that would impair the patient's ability to receive study treatment
* Other invasive malignancy within 5 years prior to Cycle 1 Day 1 except for non-invasive malignancies
* Part B : Presence of apparent radiological findings for interstitial pneumonitis or pulmonary fibrosis with pulmonary symptoms

Ages: 20 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-06-24 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2021-09-22 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse events | From the informed consent to 30 days post last dose
  Investigate the safety and tolerability of adavosertib
Incidence of Dose-limiting toxicity (DLTs) | From the first dose of Cycle 1 up to the assessment prior to the planned first dose of Cycle 2 (each cycle is 21 days for Part A and 28 days for Part B)
  Investigate the safety and tolerability of adavosertib

SECONDARY OUTCOMES:
Maximum plasma drug concentration observed (Cmax). | Part A:Samples will be collected on Cycle1Day1,5, C2D5, C3D5 and C5D5. Part B:Samples will be collected on C1D2,3 and even Cycle D2 for adavosertib and C1D1 for gemcitabine. (each cycle is 21 days for Part A, 28 days for Part B)
  PK parameters will be derived using standard, non-compartmental methods
Time of maximum plasma drug concentration observed (tmax). | Part A:Samples will be collected on Cycle1Day1,5, C2D5, C3D5 and C5D5. Part B:Samples will be collected on C1D2,3 and even Cycle D2 for adavosertib and C1D1 for gemcitabine. (each cycle is 21 days for Part A, 28 days for Part B)
  PK parameters will be derived using standard, non-compartmental methods
Area under the plasma concentration-time curve from zero to 24 hours (AUC0-24). | Part A:Samples will be collected on Cycle1Day1,5, C2D5, C3D5 and C5D5. Part B:Samples will be collected on C1D2,3 and even Cycle D2 for adavosertib and C1D1 for gemcitabine. (each cycle is 21 days for Part A, 28 days for Part B)
  PK parameters will be derived using standard, non-compartmental methods
trough plasma concentration (Ctrough). | Part A:Samples will be collected on Cycle1Day1,5, C2D5, C3D5 and C5D5. Part B:Samples will be collected on C1D2,3 and even Cycle D2 for adavosertib and C1D1 for gemcitabine. (each cycle is 21 days for Part A, 28 days for Part B)
  PK parameters will be derived using standard, non-compartmental methods
Objective response rate (ORR) | Assessed every 9 weeks in Part A and every 8 weeks in Part B with RECIST from the first dose of adavosertib until disease progression. Expected to be for up to 3 months.
  Defined as the proportion of subjects who have a best overall response of confirmed complete response (CR) or confirmed partial response (PR)
Disease control rate (DCR) | Assessed every 9 weeks in Part A and every 8 weeks in Part B with RECIST from the first dose of adavosertib until disease progression. Expected to be for up to 3 months.
  Defined as the proportion of subjects who have a best overall response of confirmed CR,confirmed PR, or stable disease (SD)
Duration of response (DoR) | Assessed every 9 weeks in Part A and every 8 weeks in Part B with RECIST from the first dose of adavosertib until disease progression. Expected to be for up to 3 months.
  Defined as the duration from the date of first documentation of response (CR or PR), which is subsequently confirmed, to the date of documented disease progression or death due to any cause in the absence of disease progression
Progressionfree free survival (PFS) | Assessed every 9 weeks with RECIST from the first dose of adavosertib until disease progression. Expected to be for up to 3 months.
  Defined as the time from the first dose of study treatment until the date of objective disease progression or death by any cause (in the absence of progression), regardless of whether the subject withdraws from the study or receives another anti-cancer therapy prior to progression
Part B: the drug interaction between adavosertib and gemcitabine. | Part B : Samples will be collected on Cycle 1 Day 2,3 and even Cycle Day 2 for adavosertib and Cycle 1 Day 1 for gemcitabine. (each cycle is 28 days)
  PK parameters will be derived using standard, non-compartmental methods

OTHER OUTCOMES:
Part B: The ctDNA samples will be analysed for predictive biomarkers of response to treatment. | Part B: at screening
  The samples may be used to develop and validate future in vitro diagnostic tests to identify patients most likely to respond to the treatment.
Part B: The ctDNA samples will be used for additional exploratory research for efficacy, tolerability, or safety assessment. | Part B: Cycle 1 Day 1 (predose), discontinuation, and progression (each cycle is 28 days).
  These samples will be used for additional exploratory research which may include but is not limited to interrogation of changes in genetic alterations associated with response or resistance to treatment as well as the dynamics of the biomarkers on treatment and potential mechanisms of resistance to treatment.
Part A: Optional exploratory biomarker research in genetic samples from subjects who have consented to participate in the genetic analysis component of the study and exploratory biomarker research for efficacy, tolerability, or safety assessment. | Part A: Cycle 1 Day 1 (each cycle is 21 days).
  To conduct potential future exploratory research into factors that may influence the progression of cancer and/or response to adavosertib.
Part B:Exploratory analyses may be undertaken on the data generated from tumour tissue to identify biomarkers of sensitivity and resistance to treatment and to increase our understanding of the disease (consenting participants only.) | Part B: at screening
  To conduct potential future exploratory research into factors that may influence the progression of cancer and/or response to adavosertib. This exploratory analysis may include immunological biomarkers such as PD-L1 expression and tumour infiltrating lymphocytes.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Chūōku, Japan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Kondo S, Katsuya Y, Yonemori K, Komuro K, Sugeno M, Kawata T, Ghiorghiu D, Meulendijks D, Yamamoto N. Safety, tolerability, pharmacokinetics, and antitumor activity of adavosertib in Japanese patients with advanced solid tumors: A phase I, open-label study. Cancer Treat Res Commun. 2024;39:100809. doi: 10.1016/j.ctarc.2024.100809. Epub 2024 Mar 24. PMID 38593512